CLINICAL TRIAL: NCT01705483
Title: A Phase 1, Multicenter, Open-Label, Dose Escalation Study of ASP9853 in Combination With Either Docetaxel or Paclitaxel in Subjects With Advanced Non-hematologic Malignancies
Brief Title: A Phase 1, Dose Escalation Study to Assess the Safety and Tolerability of ASP9853 With Either Docetaxel or Paclitaxel in Patients With Advanced Non-hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on the results of the Phase 1 data, the company decided not to pursue the development of this drug at this time.
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9853-CL-0101
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Pharmacokinetics of ASP9853; Non-hematologic Malignancies
Keywords: ASP9853; Docetaxel; Paclitaxel
MeSH Terms: interventions — ASP9853; Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1: ASP9853 with docetaxel (Experimental): 2 docetaxel dose levels and starting dose of ASP9853 followed by escalation of ASP9853 with additional dose cohorts
  Interventions: Drug: ASP9853; Drug: Docetaxel
- Part 2: ASP9853 with paclitaxel (Experimental): Starting dose for ASP9853 determined as one dose level below maximum tolerated dose (MTD) determined in Part 1, 2 paclitaxel dose levels and starting dose of ASP9853 followed by escalation of ASP9853 with additional dose cohorts
  Interventions: Drug: ASP9853; Drug: Paclitaxel

INTERVENTIONS:
Drug: ASP9853 — oral
Drug: Docetaxel — intravenous (IV)
  Other Names: Taxotere
  Arms: Part 1: ASP9853 with docetaxel
Drug: Paclitaxel — Taxol
  Other Names: intravenous (IV)
  Arms: Part 2: ASP9853 with paclitaxel

SUMMARY:
The purpose of this study is to determine the safety and tolerability and pharmacokinetics of ASP9853 combined with docetaxel or with paclitaxel in subjects with advanced non-hematologic malignancies.

DETAILED DESCRIPTION:
This is a two part study. Part 1 will test increasing dose levels of ASP9853 in combination with docetaxel. Part 2 will test increasing doses of ASP9853 combined with paclitaxel. Each part will determine the maximum tolerated dose and recommended Phase 2 dose for ASP9853 in combination with each taxane. Preliminary evidence of antitumor activity of ASP9853 in combination with docetaxel or with paclitaxel also will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a histologically or cytologically confirmed incurable, locally advanced, or metastatic non-hematologic malignancy that has progressed or failed to respond to regimens or therapies known to provide clinical benefit
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Subject must have recovered from the effects of prior systemic antineoplastic or radiation therapy(s) to ≤ Grade 1 severity or to subject's baseline values, excluding alopecia
* Subject agrees not to participate in another interventional study while on treatment

Female subject must be either:

Of non child bearing potential:

* post-menopausal (defined as at least 1 year without any menses) prior to Screening or
* documented surgically sterile or status post hysterectomy (at least 1 month prior to Screening)

Or, if of childbearing potential:

* must have a negative serum pregnancy test at Screening and
* must use two forms of birth control (at least one of which must be a barrier method) starting at Screening and throughout the study period and for 28 days after final study drug administration

Acceptable forms include:

* Established use of oral, injected or implanted hormonal methods of contraception.
* Placement of an intrauterine device (IUD) or intrauterine system (IUS).
* Barrier methods of contraception: Condom OR Occlusive cap (diaphragm or cervical/vault caps) with spermicidal
* foam/gel/film/cream/suppository
* Female subject must not donate ova starting at Screening and throughout the study period and for 28 days after final study drug administration.
* Male subject must not donate sperm starting at Screening and throughout the study period and for 28 days after final study drug administration.
* Subject with adequate bone marrow, renal, and hepatic function at baseline

Exclusion Criteria:

* Subject has received more than 3 prior cytotoxic agent-containing regimens
* Subjects with prior anaphylactic or hypersensitivity reaction to prior taxane therapy
* Subject with symptomatic central nervous system (CNS) metastases or leptomeningeal involvement
* Subjects who received treatments with any of the following:

  * Systemic chemotherapy within 21 days
  * Nitrosoureas or mitomycin C within 42 days
  * Radiotherapy to ≥ 25% of hematopoietically active bone marrow within 21 days
* Subject had major surgical procedure within 28 days or anticipates need for major surgical procedure during course of the study
* Female subjects who are breastfeeding at Screening or during the study period and for 28 days after final study drug administration.
* Subject with peripheral neuropathy > Grade 1 at baseline
* Subject with known hepatitis B surface antigen (HBsAg) positive status; or known or suspected active hepatitis C infection; or known human immunodeficiency virus (HIV) positive
* Subject with malabsorption syndrome or disease or condition significantly affecting gastrointestinal function
* Subject with significant or uncontrolled cardiac, renal, hepatic or other systemic disorders, or significant psychological conditions at baseline
* Subject with clinically significant electrocardiogram (ECG) abnormalities on 12 lead ECG performed within 14 days before start of study drug
* Subject who has received strong inhibitors or inducers of CYP3A4 within two weeks prior to start of study treatment and while on study
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half lives, whichever is longer, prior to the initiation of Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-08-28 (Actual); Primary Completion 2014-06-11 (Actual); Study Completion 2014-06-11 (Actual)

PRIMARY OUTCOMES:
Safety assessed by recording of adverse events, clinical laboratory evaluation, electrocardiograms (ECGs) physical examinations, and vital signs | Duration of study (24 months) to Final Study Visit, up to ≥ 30 days after last dose of ASP9853

SECONDARY OUTCOMES:
Pharmacokinetics (PK) Profile for ASP9853: AUC24, AUClast, AUCinf, Cmax, Ctrough, tmax, t1/2, CL/F, and Vz/F | Parts 1 and 2, Cycle 1, Day 1: Pre-dose and 9 times within the 24 hour period following ASP9853 dosing; Days 8 and 15: pre-dose, Cycles 2 + , Day 1: predose
  Area under the plasma concentration curve at 24 hours (AUC24), AUC from time zero to time of last measurable concentration (AUClast), AUC with the last concentration extrapolated to infinity (AUCinf), Maximum concentration (Cmax), Trough plasma concentration (Ctrough),Time to attain Cmax (Tmax), Apparent terminal elimination half-life (T1/2), Oral clearance (CL/F), and Volume of distribution during the terminal phase (Vz/F)
Pharmacokinetics (PK) Profile for Docetaxel: AUC24, AUClast, AUCinf, Cmax, tmax, t1/2, CL, and Vd ss | Part 1, Cycle 1, Day 1: Pre-dose and 9 times within the 24 hour period
  Clearance (CL), Distribution volume, steady state (Vd ss)
Pharmacokinetics (PK) Profile for Paclitaxel: AUC24, AUClast, AUCinf, Cmax, tmax, t1/2, CL, and Vd ss | Part 2: Cycle 1: Day 1: Pre-dose and 9 times within the 24 hour period
Objective response rate (ORR) | Treatment start to final Study Visit , up to 24 months
  The proportion of subjects with a complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) Criteria Version 1.1
Duration of response (DOR) | CR or PR response until last study visit at which a tumor assessment or an assessment of clinical disease progression is performed, up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Sarah Cannon Research Institute, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=302